CLINICAL TRIAL: NCT05522374
Title: TIRCON International NBIA (Neurodegeneration Associated With Brain Iron Accumulation) Patient Registry and Natural History Study
Brief Title: TIRCON International NBIA Registry
Acronym: TIRCON
Status: Recruiting | Type: Observational
Sponsor: LMU Klinikum (Other)
Collaborators: Seventh Framework Programme (Other); NBIA Alliance (Unknown)
Responsible Party: Principal Investigator, Prof. Thomas Klopstock, Prof. Dr. med., LMU Klinikum
Other Study IDs: TIRCON-reg
Record Dates: First submitted 2022-08-11; First posted 2022-08-31 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Neurodegeneration With Brain Iron Accumulation (NBIA); Pantothenate Kinase-associated Neurodegeneration (PKAN); Beta-Propeller Protein-Associated Neurodegeneration (BPAN); Mitochondrial Membrane Protein Associated Neurodegeneration (MPAN); Fatty Acid Hydroxylase-associated Neurodegeneration (FAHN); Kufor Rakeb Syndrome; Neuroferritinopathy; Aceruloplasminemia; Woodhouse Sakati Syndrome; COASY Protein-associated Neurodegeneration (CoPAN); PLA2G6-Associated Neurodegeneration (PLAN)
Keywords: NBIA, PKAN, BPAN, MPAN, FAHN, KRS, CoPAN, PLAN,
MeSH Terms: conditions — Pantothenate Kinase-Associated Neurodegeneration; Fatty Acid Hydroxylase-Associated Neurodegeneration; Kufor-Rakeb syndrome; Neuroferritinopathy; Familial apoceruloplasmin deficiency; Woodhouse Sakati syndrome; Neuroaxonal Dystrophies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Biospecimen Retention: Samples With DNA — RNA, DNA, Plasma and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- NBIA Patients: Patients with suspected or confirmed NBIA

SUMMARY:
TIRCON-reg aims to

* continue the provision of a global registry and natural history study for NBIA disorders
* harmonize and cover existing national and single site registries
* enable participation of countries and single sites that so far have no access to an NBIA registry
* join forces in order to recruit sufficient numbers of patients
* define the natural history of NBIA disorders
* define the most appropriate outcome measures
* inform the design and facilitate the conduction of clinical trials

DETAILED DESCRIPTION:
The TIRCON international patient registry and natural history study for patients with Neurodegeneration Associated with Brain Iron Accumulation (NBIA) was initiated and funded for the first four years by TIRCON (Treat Iron-Related Childhood-Onset Neurodegeneration), an international consortium supported by the European Union between November 1st 2011 and October 31st, 2015. Since then, the registry has been sustained through donations form Patient Organizations and industry.

Harmonization of existing data has been performed by establishing and applying matching and transformation rules. The web-based registry is now fully functional for a critically needed natural history study of all NBIA subtypes. A focus has been set on scores that are most appropriate to reflect stage and progression of disease, e.g. the Barry Albright Dystonia scale, the Patient´s Global Impression of Improvement (PGII), the Unified Parkinson Disease Rating Scale (UPDRS; parts I-III and VI) and quality-of-life scores. The natural history data are collected yearly, or in rapidly progressing cases every six months, if applicable. Patients who present to one of our centers are eligible after informed consent to participate.

ELIGIBILITY:
Inclusion Criteria:

* suspected or confirmed NBIA
* willingness to participate

Exclusion Criteria:

* unwillingness to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: children, adults, patients with limited decision-making capacity
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2012-06-14 (Actual); Primary Completion 2040-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
Change in Score on the Barry-Albright Dystonia (BAD) Scale | The individual participants are followed with annual assessments over a long time period (up to 30 years) or until discontinuation or death.
  The Barry-Albright Dystonia Scale is an instrument for rating the severity of dystonia in eight body regions. The individual scores are summed to provide a total score that ranges from 0 to 32; the higher the score, the more severe the dystonia. Patients with dystonia are assessed for the change in total BAD score over time since Baseline.
Change in Score on Unified Parkinson's Disease Rating (UPDRS) Scale, Part I-III, VI | The individual participants are followed with annual assessments over a long time period (up to 30 years) or until discontinuation or death.
  The Unified Parkinson's Disease Rating Scale (UPDRS) is the major rating scale used to assess severity of symptoms of Parkinson's disease, some of which are similar to symptoms in NBIA. The UPDRS subscales used in this study are Part I: Mentation, Behavior and Mood, scored from 0 (best) to 16 (worst); Part II: Activities of Daily Living, scored from 0 (best) to 52 (worst); Part III: Motor Examination, scored from 0 (best) to 108 (worst); and Part VI: Schwab and England Activities of Daily Living Scale, scored from 0% (worst) to 100% (best).
Change in Score on Pediatric Quality of Life (PedsQL) | The individual participants are followed with annual assessments over a long time period (up to 30 years) or until discontinuation or death.
  The Pediatric Quality of Life (PedsQL) questionnaire is used to measure functional health and well-being from the patient's point of view. Separate versions of the questionnaire are available for children, young adults aged 18-25 years, and adults older than 25 years. Patients are asked to indicate how they have felt over the past month, and the scores of the 23 questions are used to generate an overall score that ranges from 0 (worst) to 100 (best).
Disease progression | The individual participants are followed with annual assessments over a long time period (up to 30 years) or until discontinuation or death.
  Disease progression as assessed by clinical examination and captured as HPO (Human Phenotype Ontology) Terms at each visit.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Klopstock, Prof. Dr., Principal Investigator — LMU Klinikum, Friedrich-Baur-Institute
Locations (9):
- Children's Hospital of Eastern Ontario, Division of Neurology, Department of Pediatrics, Ottawa, Canada
- Charles University, Department of neurology, Prague, Czechia
- LMU Klinikum, Friedrich-Baur-Institute, Munich, Bavaria, Germany
- The Foundation of the Carlo Besta Neurological Institute, IRCCS, Milan, Italy
- University medical Center Groningen (UMCG) Department of Neurology AB 51, Groningen, Netherlands
- The Childrens Memorial Health Institute, Warsaw, Poland
- University of Belgrade, Department of Movement Disorders and Degenerative Brain Diseases, Belgrade, Serbia
- Spain (2):
  - Hospital Vall d'Hebron - Institut de Recerca (VHIR), Pediatric Neurology, Movement Disorders, Barcelona
  - Hospital Sant Joan de Déu, Universitat de Barcelona, Servei de Neurología, Barcelona

IPD SHARING:
Plan to Share IPD: Yes
Any data or requests from the project can be shared with researchers upon written request. Data sharing requires i) the approval by the respective scientific committee and ii) an approval by the institutional review board of the researcher on the intended project.
Supporting Information: ICF
Time Frame: ime frame for data usage needs to be specified in the proposal for data sharing
Access Criteria: Approved written proposal including description of the research plan and data usage purpose.

REFERENCES:
- [Background] Kalman B, Lautenschlaeger R, Kohlmayer F, Buchner B, Kmiec T, Klopstock T, Kuhn KA. An international registry for neurodegeneration with brain iron accumulation. Orphanet J Rare Dis. 2012 Sep 17;7:66. doi: 10.1186/1750-1172-7-66. PMID 22985983
- [Background] Klopstock T, Tricta F, Neumayr L, Karin I, Zorzi G, Fradette C, Kmiec T, Buchner B, Steele HE, Horvath R, Chinnery PF, Basu A, Kupper C, Neuhofer C, Kalman B, Dusek P, Yapici Z, Wilson I, Zhao F, Zibordi F, Nardocci N, Aguilar C, Hayflick SJ, Spino M, Blamire AM, Hogarth P, Vichinsky E. Safety and efficacy of deferiprone for pantothenate kinase-associated neurodegeneration: a randomised, double-blind, controlled trial and an open-label extension study. Lancet Neurol. 2019 Jul;18(7):631-642. doi: 10.1016/S1474-4422(19)30142-5. PMID 31202468
- [Background] Karin I, Buchner B, Gauzy F, Klucken A, Klopstock T. Treat Iron-Related Childhood-Onset Neurodegeneration (TIRCON)-An International Network on Care and Research for Patients With Neurodegeneration With Brain Iron Accumulation (NBIA). Front Neurol. 2021 Feb 22;12:642228. doi: 10.3389/fneur.2021.642228. eCollection 2021. PMID 33692746
- [Background] Iankova V, Karin I, Klopstock T, Schneider SA. Emerging Disease-Modifying Therapies in Neurodegeneration With Brain Iron Accumulation (NBIA) Disorders. Front Neurol. 2021 Apr 15;12:629414. doi: 10.3389/fneur.2021.629414. eCollection 2021. PMID 33935938
- See also: Project website — http://tircon.eu